CLINICAL TRIAL: NCT05299697
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Study of TG103 Injection in the Management of Overweight or Obesity
Brief Title: A Study of TG103 Injection in Overweight or Obesity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSA1803-007
Record Dates: First submitted 2022-03-03; First posted 2022-03-29 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TG103 15 mg (Experimental): Administered subcutaneously (s.c., under the skin) once every week for 24 weeks. Doses gradually increased to 15 mg.
  Interventions: Drug: TG103 15 mg
- TG103 22.5 mg (Experimental): Administered subcutaneously (s.c., under the skin) once every week for 24 weeks. Doses gradually increased to 22.5 mg.
  Interventions: Drug: TG103 22.5 mg
- Placebo (Placebo Comparator): Administered subcutaneously (s.c., under the skin) once every week for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TG103 15 mg — Administered subcutaneously (s.c., under the skin) as well as calorie restrict diet and increased physical activity for 24 weeks. Doses gradually increased from 7.5 mg to 15 mg.
  Arms: TG103 15 mg
Drug: TG103 22.5 mg — Administered subcutaneously (s.c., under the skin) as well as calorie restrict diet and increased physical activity for 24 weeks. Doses gradually increased from 7.5 mg, 15 mg to 22.5 mg.
  Arms: TG103 22.5 mg
Drug: Placebo — Administered subcutaneously (s.c., under the skin) as well as calorie restrict diet and increased physical activity for 24 weeks.
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled, parallel phase II study to evaluate efficacy, safety, pharmacokinetics characteristics and immunogenicity of two dose levels of TG103 injection, a GLP-1 receptor agonist, in the management of overweight or obesity, to support dose selection for further development.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years ≤ age ≤ 75 years.
* Body Mass Index (BMI) ≥ 28 kg/m^2, or 24 kg/m^2 < BMI ≤ 28 kg/m^2 with at least one of obesity-related complications.
* Regular diet and exercise and stable body weight (i.e. <5 kg self-reported change) within 12 weeks before screening as well as body weight ≥ 60 kg at screening.
* Weight loss less than 5% or weight increase after simple diet and exercise efforts for at least 3 months.
* Be able to understand the trial and complete the procedures, and be voluntary to participate in this study and sign the informed consent.

Exclusion Criteria:

* Screening HbA1c ≥ 6.5%, or screening FPG ≥ 7.0mmol/L or<2.8mmol/L, or history of diabetes mellitus or hypoglycemia.
* Overweight or obesity due to single gene mutation, disease or drug, or weight increase due to non-fat mass increase.
* Treatment with any medication or product which in the investigator's opinion will cause change in weight to influence trial evaluations within 12 weeks before screening or during this study.
* Subjects who underwent bariatric surgery within 12 months before screening, or are not yet recovered from any surgery or injury at screening.
* Subjects who participated in any clinical trial and received the treatment within 12 weeks before screening, or who participated in the clinical trial and received treatment with TG103 injection.
* History of allergy or suspected allergy to GLP-1 receptor agonists or antibody agents, or other severe allergy history based on which the subjects may be allergic to the study drugs in investigator's opinion.
* Personal history or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2 (MEN-2), or screening calcitonin ≥ 50 ng/L.
* Previous history or screening ultrasound includes one of the following: chronic pancreatitis, acute pancreatitis, gallstone with at least one of less than 5mm, choledocholithiasis, except that there was no cholelithiasis after treatment or cholecystectomy.
* No recovery from gastrointestinal disease or symptom at screening, or previous withdrawl of GLP-1 receptor agonist, GLP-1/GIP receptor agonist, GLP-1/GCG receptor agonist or metformin by gastrointestinal adverse drug reaction, or previous history of gastrointestinal surgery that influences the gastrointestinal motility in the investigators' opinions.
* Acute infection at screening.
* History of easily relapsed skin disease (e.g. urticaria), or present skin injury in any administration site at screening.
* History of acute coronary syndrome, stroke, severe asthma, epilepsy, systemic lupus erythematosus, hemolytic anemia, cirrhosis and the other severe disease, or history of malignant tumor.
* One of the followings at screening: systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg, or NYHA ≥ grade III, or QTc interval prolongation (i.e. QTcF>450ms in males or >470ms in females) or severe arrhythmia (e.g. atrioventricular block equal to or more than II degree, ventricular tachycardia).
* History of abnormal thyroid function with requirement of medication treatment at screening, or TSH beyond the normal reference range at screening.
* One of the followings at screening: 1) ALT or AST>3 × UNL (upper normal limit), or total bilirubin>1.5 × UNL, 2) blood amylase or lipase>1.5 × UNL, 3) TG>5.6mmol/L, 4) eGFR<60ml/min/1.73m^2 (calculated by CKD-EPI formula), 5) HBsAg, HCV-antibody, HIV-antibody or anti-TP antibody positive, 6) WBC< 3×10^9/L, or Hb <100g/L, 7) INR>1.2.
* History of drug abuse, drug dependence or alcoholism.
* History of moderate to severe depression, or screening Patient Health Questionaire-9 (PHQ-9) score ≥ 15.
* The fertile female who is pregnant, breast-feeding or with blood HCG positive at screening, or the fertile male or female cannot use an effective contraceptive method during the trial and for 3 months after the end of treatment.
* Other situations that are not suitable for the study in the investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Relative change from baseline in body weight at week 24 | From baseline to week 24
  percent change in body weight

SECONDARY OUTCOMES:
Relative change from baseline in body weight (%) at week 12 and week 27 | From baseline to week 27
  percent change in body weight
Proportion of subjects with weight loss of ≥ 5% and ≥ 10% of baseline body weight at week 12 and week 24 | From baseline to week 24
Change from baseline to 12 weeks, 24 weeks and 27 weeks in body weight | From baseline to week 27
  weight in kg
Change from baseline to 12 weeks, 24 weeks and 27 weeks in BMI | From baseline to week 27
  BMI in kg/m^2
Change from baseline to 12 weeks, 24 weeks and 27 weeks in waist to hip circumference ratio | From baseline to week 27
  waist circumference and hip circumference will be combined to report waist to hip circumference ratio
Change from baseline to 12 weeks, 24 weeks and 27 weeks in waist circumference | From baseline to week 27
  waist circumference in cm
Change from baseline to 12 weeks and 24 weeks in HbA1c | From baseline to week 24
  HbA1c in %
Change from baseline to 12 weeks and 24 weeks in FPG (fasting plasma glucose) | From baseline to week 24
  FPG (fasting plasma glucose) in mmol/L
Change from baseline to 12 weeks and 24 weeks in FINS (fasting insulin) | From baseline to week 24
  FINS (fasting insulin) in mU/L
Change from baseline to 12 weeks and 24 weeks in fasting C peptide | From baseline to week 24
  fasting C peptide in nmol/L
Change from baseline to 12 weeks and 24 weeks in HOMA-IR | From baseline to week 24
  FPG and FINS will be combined to report HOMA-IR in mmol/mU
Change from baseline to 12 weeks and 24 weeks in TC（total cholesterol） | From baseline to week 24
  TC in mmol/L
Change from baseline to 12 weeks and 24 weeks in TG（triglyceride） | From baseline to week 24
  TG in mmol/L
Change from baseline to 12 weeks and 24 weeks in LDLC（low density lipoprotein cholesterol） | From baseline to week 24
  LDLC in mmol/L
Change from baseline to 12 weeks and 24 weeks in HDLC（high density lipoprotein cholesterol） | From baseline to week 24
  HDLC in mmol/L
Change from baseline to 12 weeks and 24 weeks in systolic blood pressure and diastolic blood pressure | From baseline to week 24
  systolic blood pressure, diastolic blood pressure in mmHg, respectively
Change from baseline to 12 weeks and 24 weeks in scores of the patient health questionnaire (PHQ-9) | From baseline to week 24
  There are 9 items in PHQ-9 and the score ranges from 0-3 for each item. The total score will be the sum of the scores of all items.
Number of TEAEs and SAEs from baseline to week 27 | From baseline to week 27

OTHER OUTCOMES:
Ctrough (the trough plasma concentration of TG103) | From baseline to week 24
  Ctrough will be measured once every 4 week until week 24.
Number of participants with Anti-TG103 antibodies positive | From baseline to week 27
  Anti-TG103 antibodies will be measured once every 4 week until week 27.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Baotou City Central Hospital, Baotou, Neimenggu, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.